CLINICAL TRIAL: NCT03966196
Title: Validation and Characterization of Signal Decrease on an Oximeter in Chronic Obstructive Pulmonary Disease
Brief Title: Validation and Characterization of Signal Decrease on an Oximeter in COPD (They Have Chronic Obstructive Pulmonary Disease) Patients During Deep Inhalation (
Acronym: OXYMETRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/25AVR/185
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Disease; Copd
Keywords: COPD
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: half healthy subject, half COPD patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Other): oxymetry and finger pressure in Healthy subjects
  Interventions: Other: Measurements of oxygen saturation and finger pressure during deep inspiration
- COPD patients (Experimental): oxymetry and finger pressure in COPD patients
  Interventions: Other: Measurements of oxygen saturation and finger pressure during deep inspiration

INTERVENTIONS:
Other: Measurements of oxygen saturation and finger pressure during deep inspiration — Measurements during deep inspiration of oxygen saturation with pulse oximeter and finger pressure with pressure cuff

SUMMARY:
The objective is to verify that there is a decrease in the pulsed oxygen saturation with the digital sensor. That is, the drop in oxygen saturation in COPD patients during inhalation is real and not due to an artifact of the measuring tool, because oximeters need a quality pulsatile signal to properly measure oxygen saturation

ELIGIBILITY:
healthy arm

Inclusion Criteria:

* Healthy adults volunteers are recruited from students with normal lung function.

Exclusion Criteria:

* abnormal lung function

COPD Arm

Inclusion Criteria:

* Adults with Chronic Obstructive pulmonary disease

Exclusion Criteria:

* cardiovascular disease

The subjects selected are selected on a voluntary basis among the patients coming to the pulmonary consultation. They have Chronic Obstructive Pulmonary Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
drop in oxygen saturation during deep inspiration in COPD | from the intervention to 3 minutes after the start of the intervention
  saturation is measured in percentage (SPO2)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Liistro, PhD, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No